CLINICAL TRIAL: NCT04501133
Title: Sensory-specific Peripheral Stimulation for Tremor Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Jose Pons, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU00211930
Record Dates: First submitted 2020-07-21; First posted 2020-08-06 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease; Essential Tremor
Keywords: Parkinson's Disease; Essential Tremor; Peripheral electrical stimulation; Transcranial magnetic stimulation; High-density electromyography; Electroencephalography; Magnetic resonance imaging
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to understand how motor activation can be reduced. For this purpose, it will be examined how some muscles of the arm respond to electric and magnetic stimulation. The effects of the electric and/or magnetic stimulation will be recorded non-invasively with HD-EMG.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Participants (Experimental): Healthy participants without motor disorders and medications influencing brain functions will be scanned with MRI and undergo PES and/or single pulse TMS during several visits, each with different stimulation patterns, while HD-EMG is recorded.
  Interventions: Device: Peripheral electrical stimulation; Device: Single pulse TMS
- Patients (Experimental): Participants with Parkinson's Disease or essential tremor will be scanned with MRI and undergo PES and/or single pulse TMS during several visits, each with different stimulation patterns, while HD-EMG and EEG are recorded.
  Interventions: Device: Peripheral electrical stimulation; Device: Single pulse TMS

INTERVENTIONS:
Device: Peripheral electrical stimulation — Electrical stimulation will be delivered to forearm muscles with an electrical stimulator (Digitimer Ltd., Hertfordshire, UK) so that they generate forces opposed to those arising from the tremorgenic input.
Device: Single pulse TMS — Single-pulse TMS (spTMS) will be delivered with a TMS stimulator (MagPro X100 w/ MagOption, MagVenture, Farum, Denmark) and a figure-of-eight TMS coil. An MRI-based TMS navigation system will be used to navigate the TMS coil (Localite, St Augustin, Germany).

SUMMARY:
The purpose of this study is to understand the neurophysiological mechanisms of peripheral electrical stimulation (PES) in modulating supraspinal tremorogenic input to motoneurons. For this purpose, the investigators will use transcutaneous PES, high-density electromyography (HD-EMG), transcranial magnetic stimulation (TMS), electroencephalography (EEG), magnetic resonance imaging (MRI), and neuromusculoskeletal modelling. This study will be carried out in both healthy participants and patients with essential tremor (ET) and Parkinson's disease (PD).

DETAILED DESCRIPTION:
In Experiment A, the investigators will recruit healthy participants without motor disorders and medications influencing brain function (n = 25). The investigators will characterize inhibition of wrist flexors/wrist extensors and first dorsal interossei (FDI) and abductor pollicis brevis (APB) muscles with PES, and also use TMS to stimulate the corresponding areas in the brain and see if the movement can be reduced through PES. HD-EMG will be used to collect data and identify associated motor unit spike trains. Motor-evoked potentials (MEPs) will be recorded with EMG when TMS is targeted to the primary motor cortex. Resting state functional magnetic imaging resonance (rs-fMRI) and high-angular resolution diffusion imaging (HARDI) tractography of the brain will be recorded.

In Experiment B, the investigators will recruit patients with essential tremor (ET) and/or Parkinson's disease (PD) (n = 25 for each pathology). The investigators will repeat the same characterization of inhibition of wrist flexors/wrist extensors and PDI/APB with PES and also use TMS to stimulate corresponding areas in the brain. Additionally, the investigators will test PES conditions as a tremor reduction strategy at the wrist level. The investigators will also test PES conditions at the elbow and shoulder joints as a tremor reduction strategy. Finally, the investigators will observe and characterize the long-term effects (lasting 24h, 48h, and 7 days post stimulation) of PES via coherence between HD-EMG and EEG at the tremor frequency.

ELIGIBILITY:
Inclusion Criteria for Healthy Participants:

* Age from 18 to 80 years
* No history of a brain and/or skull lesion
* Normal hearing and (corrected) vision
* Able to understand and give informed consent
* No neurological disorders, no tremor
* Absence of pathology that could cause abnormal movements of extremities (e.g., epilepsy, stroke, marked arthritis)
* Able to understand and speak English

Inclusion Criteria for Patients:

* Age from 18 to 80 years
* No prior history of skull lesions or craniotomy
* Normal hearing and (corrected) vision
* Able to understand and give informed consent
* Diagnosis of ET (Tremor Research investigation Group criteria) or diagnosis of PD (UK PD Society Brain bank diagnostic criteria) by a physician
* Tremor in at least an upper limb with pure flexion-extension wrist tremor with posture (ET) and rest (PD).
* Tremor at least moderate-severe by clinician judgment and tremor scales (Fahn Tolosa Marin Tremor Rating Scale (TETRAS), Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS))
* Absence of pathology that could cause abnormal movements of extremities (e.g., epilepsy, stroke, marked arthritis, moderate to severe dyskinesias in PD)
* Stable medication doses for at least 30 days prior to study enrollment
* Able to understand and speak English

Exclusion Criteria for Healthy Participants:

* Cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps
* Metal in the body (rods, plates, screws, shrapnel, dentures, IUD) or metallic particles in the eye
* Surgical clips in the head or previous neurosurgery
* Any magnetic particles in the body
* Cochlear implants
* Prosthetic heart valves
* Epilepsy or any other type of seizure history
* Any neurological diagnoses or medications influencing brain function
* History of significant head trauma (i.e., extended loss of consciousness, neurological sequelae)
* Known structural brain lesion
* Significant other disease (heart disease, malignant tumors, mental disorders)
* Significant claustrophobia; Ménière's disease
* Pregnancy (ruled out by urine ß-HCG if answers to screening questions suggest that pregnancy is possible), breast feeding
* Non prescribed drug use
* History of current substance abuse (exception: current nicotine use is allowed)
* Recreational marijuana
* Tremor, parkinsonism; neurological diseases; medical (cardiological, renal, hepatic, oncological) or psychiatric disease that would interfere with study procedures for asES, HD-EMG, TMS, or EEG
* Dementia; severe depression; or prior neurosurgical procedures
* Failure to perform the behavioral tasks or neuropsychological evaluation tests
* Prisoners

Exclusion Criteria for Patients:

* Cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps
* Metal in the body (rods, plates, screws, shrapnel, dentures, IUD) or metallic particles in the eye
* Surgical clips or shunts in the head
* Any magnetic particles in the body
* Cochlear implants
* Prosthetic heart valves
* Epilepsy or any other type of seizure history
* Significant claustrophobia; Ménière's disease
* Pregnancy, breast feeding
* Medications increasing risk for seizures
* History of current substance abuse (exception: current nicotine use is allowed)
* Failure to perform tasks (e.g., follow instructions to stay still in the scanner) or fill in safety screening forms
* Prisoners
* Atypical or secondary parkinsonism
* Co-existence of other neurological diseases
* Mixed or complex tremors
* Inability or unwillingness to discontinue medications for tremor on the day of study assessments
* Medical (cardiological, renal, hepatic, oncological) or psychiatric disease that would interfere with study procedures for asES, HD-EMG, TMS, or EEG; dementia; severe depression; prior neurosurgical procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Amount of Motor Inhibition | Experiment A: Short-term: before vs. during and at 1 minute after PES. Experiment B: Short-term: before vs. during and at 1 minute after PES. Long-term: persistence of changes at post 24 hours, post 48 hours, and post 1 week after PES.
  HD-EMG will be recorded with a 64-channel device (EMG-Quattrocento; 400-channel EMG amplifier, OT Bioelettronica, Italy). The HD-EMG data will be recorded at the wrist level before, during and after muscle contractions. All data will be analyzed offline. Changes in the amount of inhibition will be assessed. The amount of inhibition is calculated as the mean discharge rate across trials and normalized as a percentage of the baseline (100%). To assess the short-term effects, HD-EMG data will be collected before (baseline), during and 1 minute (Post) after PES. Changes in amount of motor inhibition will be measured by comparing the amount of inhibition before (baseline), during and 1 minute after PES (Post). To assess long-term effects, HD-EMG data will be collected at post 24h, post 48h, and post 1 week after PES. The amount of inhibition at 24h, 48h, and 1 week after PES will be compared with the baseline amount of inhibition (before PES).
Changes in motor evoked potentials (MEPs) | Experiment A: Short-term: before vs. during and at 5 minutes after PES. Experiment B: Short-term: before vs. during and at 5 minutes after PES. Long-term: persistence of changes at post 24 hours, post 48 hours, and post 1 week after PES.
  To assess the effects of electrical stimulation in motor inhibition, single-pulse TMS will be administered to the contralateral area of the brain while MEPs are recorded from the contralateral site (EMG-Quattrocento; 400-channel EMG amplifier, OT Bioelettronica, Italy). The mean peak-to peak MEP amplitude will be calculated to assess changes in inhibition. To assess the short-term effects, MEP data will be collected before (baseline), during and 5 minutes (Post) after PES. Changes in MEPs will be measured by comparing the MEPs before (baseline), during and 1 minute after PES (Post). To assess long-term effects, MEP data will be collected at post 24h, post 48h, and post 1 week after PES. The MEPs at 24h, 48h, and 1 week after PES will be compared with the baseline MEPs (before PES).
Changes in cortico-muscular coherence in ET and/or PD participants | Experiment A: N/A. Experiment B: Short-term effects, within sessions (before vs. 1 minute after PES. Long-term effects, across sessions (persistence of changes at post 24 hours, post 48 hours, and post 1 week after PES).
  EEG will be recorded with a 64-channel whole-head device (NeurOne, Bittium, Kuopio, Finland) and HD-EMG with a 64-channels system (EMG-Quattrocento; 400-channel EMG amplifier, OT Bioelettronica, Italy). The coherence between EEG and HD-EMG signals will be computed to assess supraspinal and spinal inhibition. To assess the short- term effects, EEG and HD-EMG data will be collected before (Pre) and 1 minute (Post) after PES. Changes in cortico-muscular coherence will be measured by comparing the cortico-muscular coherence before (baseline) and 1 minute after PES (Post). To assess long-term effects, EEG and HD-EMG data will be collected at post 24h, post 48h, and post 1 week after PES. The cortico-muscular coherence at 24h, 48h, and 1 week after PES will be compared with the baseline cortico-muscular coherence (before PES).
Changes in kinematics | Experiment A: N/A. Experiment B: Short-term effects, within sessions (before vs. 1 minute after PES). Long-term effects, across sessions (persistence of changes at post 24 hours, post 48 hours, and post 1 week after PES).
  Tremor amplitude will be measured with inertial measurement units that quantify variations in wrist angles during tremor. Specifically, the tremor amplitude will be calculated as the mean peak-to-peak amplitude between maximal wrist flexion and wrist extension angles. To assess the short-term effects, tremor amplitude will be collected before (Pre) and 1 minute (Post) after PES. Changes in tremor amplitude will be measured by comparing the tremor amplitude before (baseline) and 1 minute after PES (Post). To assess long-term effects, tremor amplitude will be recorded at post 24h, post 48h, and post 1 week after PES. The tremor amplitude at 24h, 48h, and 1 week after PES will be compared with the baseline tremor amplitude (before PES).

SECONDARY OUTCOMES:
Clinical motor score change | For Experiment A: N/A. For Experiment B: Short-term effects, within sessions (before and after PES). Long-term effects, across sessions (persistence of changes at 24 hours, 48 hours, and 1-week after PES).
  The MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and the Fahn Tolosa Marin (FTM) rating scale are functional scales used by clinicians to assess the functional impairments caused by Parkinson's disease and essential tremor, respectively. The MDS-UPDRS and the FTM scales will be used to assess clinical motor changes induced by the PES. To assess the short-term effects, The MDS-UPDRS or the FTM will be administered before and after PES. Changes in scores will be assessed by comparing the MDS-UPDRS/or FTM scores before (baseline) and after PES (Post). To assess long-term effects, the MDS-UPDRS/or FTM scores will be collected at post 24h, post 48h, and post 1 week after PES. The MDS-UPDRS/or FTM scores at 24h, 48h, and 1 week after PES will be compared with the baseline the MDS-UPDRS/or FTM scores (before PES).
MRI/rs-fMRI connectivity | Experiment A: Baseline and through study completion, an average of 3 months. Experiment B: Baseline and through study completion, an average of 6 months.
  Structural connectivity will be assessed with diffusion tensor imaging (DTI). Functional connectivity will be assessed with resting-state MRI (rs-MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Pons, Ph.D, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pascual-Valdunciel A, Kurukuti NM, Montero-Pardo C, Barroso FO, Pons JL. Modulation of spinal circuits following phase-dependent electrical stimulation of afferent pathways. J Neural Eng. 2023 Jan 27;20(1). doi: 10.1088/1741-2552/acb087. PMID 36603216